CLINICAL TRIAL: NCT02432001
Title: Radiologically Guided Biopsies of Metastatic Castration Resistant Prostate Cancer (mCRPC) to Identify Adaptive Mechanisms of Resistance
Brief Title: Radiologically Guided Biopsies of mCRPC
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: American Association for Cancer Research (Other)
Responsible Party: Sponsor
Other Study IDs: 125519
Record Dates: First submitted 2015-04-28; First posted 2015-05-01 (Estimated); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Image-Guided Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Image-Guided Biopsies: Image-guided biopsies will be performed at the Dream Team Site enrolling the patient. Lesions will be chosen based upon the strength of the evidence suggesting the presence of metastasis and with the goal of minimizing patient risk. Soft tissue lesions and lesions with documented radiologic progression should be prioritized for biopsy. If the Radiologist in charge of the procedure cannot identify a lesion amenable for biopsy, the patient will be considered a screening failure.
  Interventions: Procedure: Image-Guided Biopsies

INTERVENTIONS:
Procedure: Image-Guided Biopsies

SUMMARY:
The purpose of this study is to better understand how cancer treatment may affect cancer cells. The research will involve genetic, molecular, cellular, and immunologic experiments using blood and tumor specimens. It is hoped that the information gained from these studies will lead to a greater understanding of castrate-resistant prostate cancer and potentially, improvements in cancer treatment.

This is a tissue collection protocol requiring image-guided biopsies of metastatic, castration-resistant prostate cancer (mCRPC). The investigators will focus on enrolling patients with metastatic CRPC who have progressed while receiving novel AR-targeted therapeutics such as abiraterone and enzalutamide. This population of patients was selected because resistance develops relatively rapidly following potent inhibitors of AR activity and the mechanisms of resistance have to be better understood. Without comprehensive analysis of mCRPC tumor, the investigators will never gain a full understanding of the biology driving resistance in human disease and developing rational co-targeting approaches will not be possible.

ELIGIBILITY:
Inclusion Criteria:

* History of histologically confirmed prostate cancer. Patients without histologically confirmed prostate cancer are eligible if both the treating physician and the study investigator agree that the patient's history is unambiguously indicative of advanced prostate cancer (e.g. high PSA responsive to Androgen Deprivation Therapy.)
* Radiographic evidence of metastatic disease amenable to image-guided biopsy of a metastatic site. Soft-tissue as well as bony metastatic lesions will be considered acceptable. Patients with locally advanced disease only (where the biopsy would be of a prostatic mass) are not eligible. Biopsy of newly emerging radiographic metastases is desired and preferable to the biopsy of previously existing lesions whenever possible.
* Platelets >75,000/μl within 14 days prior to biopsy
* Prothrombin time (PT) or International Normalized Ratio (INR) and a partial thromboplastin time (PTT) < 1.5 times the institutional upper limit of normal (ULN) within 14 days prior to biopsy.
* Patients on warfarin, aspirin, or other anti-coagulants are eligible provided they are deemed able to tolerate discontinuation of anti-coagulation for one week prior to the biopsy. Conversion to low molecular weight heparin prior to biopsy is permitted per local standard operating procedures, provided there is agreement regarding the procedure between the treating physician, the interventional radiologist and the PI.
* Castrate levels of testosterone (testosterone <50n g/dL) within 28 days prior to biopsy.
* Patients with significant congenital or acquired bleeding disorders (eg von Wildebrand's disease, acquired bleeding factor inhibitors) are not eligible.
* If no prior orchiectomy, medical castration therapy must continue while on study.
* Prostate-specific antigen (PSA) level obtained within 28 days prior to biopsy.
* Patients currently on first generation oral anti-androgens (flutamide, bicalutamide, nilutamide) must have progressed after at least 4 weeks of anti-androgen discontinuation.
* Patient's disease is currently progressing (in setting of testosterone < 50 ng/dl), defined by any of the following criteria:
* PSA Progression: PSA level of at least 2 ng/ml which has risen on at least 2 successive occasions, at least one week apart. If the confirmatory PSA (#3) value is less (i.e., #3b) than the screening PSA (#2) value, then an additional test for rising PSA (#4) will be required to document progression for the purposes of eligibility.
* Soft tissue progression: by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Bone scan progression: the appearance of >=2 new lesions. Symptomatic progression in an area of radiologically evident disease.
* One of the following criteria must be met:
* Evidence of disease progression (as defined above) following treatment with at least 2 months of abiraterone acetate, enzalutamide, or ARN509 - based therapy.
* Enrollment on a high priority clinical trial conducted by the West Coast Dream Team (WCDT). Examples include trials with biopsy obtained before abiraterone or enzalutamide therapy, and following development of resistance to those agent(s). This list is maintained by the lead site.
* Evidence of disease progression (as defined above) in patients with "aggressive phenotype" metastatic castration resistant prostate cancer (mCRPC) with at least one of the following clinical features
* Visceral or brain metastases
* Known small cell or neuro-endocrine subtypes (by Immunohistochemistry (IHC) or serum markers)
* Primary androgen deprivation therapy (ADT) resistance defined as a nadir PSA of > 4 ng/dl after 7 months of primary androgen deprivation (with Testosterone < 50 ng/dl.)
* Prior chemotherapy for Castration Resistant Prostate Cancer is not allowed
* Age > 18 years
* Eastern Cooperative Oncology Group (ECOG) Performance status 0-3
* Ability to understand and the willingness to sign a written informed consent document

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prostate Cancer
Sampling Method: Non-Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2013-02-22 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Proportion of mCRPC patients with high androgen receptor activity | Up to 2 years
  Determined by a gene-expression-based signature for Androgen Receptor activity having a probability of >0.50

SECONDARY OUTCOMES:
Progression Free Survival | Up to 2 years
  Measured from the start of therapy after the baseline biopsy until progression. Patients not progressing will be censored at the date of last clinical follow-up or date of last contact, respectively.
Overall Survival | Up to 2 years
  Measured from the start of therapy after the baseline biopsy until death. Patients not progressing or dying will be censored at the date of last clinical follow-up or date of last contact, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Eric Small, MD, Principal Investigator — University of California, San Francisco
Locations (5):
- United States (4):
  - University of California, Davis, Davis, California
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Francisco, California
  - Oregon Health & Science University, Portland, Oregon
- University of British Columbia, Vancouver, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aggarwal R, Huang J, Alumkal JJ, Zhang L, Feng FY, Thomas GV, Weinstein AS, Friedl V, Zhang C, Witte ON, Lloyd P, Gleave M, Evans CP, Youngren J, Beer TM, Rettig M, Wong CK, True L, Foye A, Playdle D, Ryan CJ, Lara P, Chi KN, Uzunangelov V, Sokolov A, Newton Y, Beltran H, Demichelis F, Rubin MA, Stuart JM, Small EJ. Clinical and Genomic Characterization of Treatment-Emergent Small-Cell Neuroendocrine Prostate Cancer: A Multi-institutional Prospective Study. J Clin Oncol. 2018 Aug 20;36(24):2492-2503. doi: 10.1200/JCO.2017.77.6880. Epub 2018 Jul 9. PMID 29985747